CLINICAL TRIAL: NCT06638073
Title: Continuous Connected Patient Care (CCPC), a Pilot Testing a Novel Device for Continuous Vitals Monitoring - Department of Anesthesia at PHC
Status: Recruiting | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Collaborators: Excelar (Unknown); Cloud DX Inc. (Industry); Bridge Health Solutions (Unknown); Providence Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: H24-00862
Record Dates: First submitted 2024-09-16; First posted 2024-10-15 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Surgical Procedure, Unspecified; Intensive Care Units (ICUs)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To confirm feasibility and accessibility of the CCPC Platform (Oxymotion, Bridge Health Solutions medication adherence software, CloudDX home kit) in two different environments - in hospital and at-home, in patients undergoing non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* Patients that have undergone a non-cardiac surgery at SPH requiring an inpatient hospital stay
* Peri-op patients who are in the Surgical High Acuity Unit (SHAU) and those followed by Anesthesia Perioperative Outreach team on the ward
* Living within British Columbia, Canada and in an area that is covered by Bell cellular network

Exclusion Criteria:

* Patient refusal
* Lack of capacity to consent to the study (including having received sedative or general anesthetic within the past 24 hours)
* Unable to use (or does not have a caregiver who can help put on) study monitoring device at home
* Unable to complete (or does not have a caregiver who can help complete) study questionnaires by electronic (mobile, tablet, or computer), paper, nor phone
* No access to cell phone nor landline at home to receive follow-ups
* Preoperatively known to be discharged to a nursing home or rehabilitation facility
* Known allergic reactions to any part material of study devices

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have undergone a non-cardiac surgery requiring an inpatient hospital stay and peri-op patients who are in the Surgical High Acuity Unit (SHAU) at SPH.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Collect patient and clinicians' feedback about the CCPC Platform | From enrollment to the end of follow up at 10 days
  This will be completed via an assessment of the quantitative data on how long and how often patients use this monitoring and what were the reasons that patients took the monitors on and off.
Confirm the technical goals of the CCPC platform are met. | From enrollment to the end of follow up at 10 days
  This will be completed by ensuring clinical workflow is met when using the monitoring platform.
Collect patient and clinicians' feedback about the CCPC Platform | From enrollment to the end of follow up at 10 days
  This will be completed via an assessment of the Usability questionnaires.
Collect patient and clinicians' feedback about the CCPC Platform | From enrollment to the end of follow up at 10 days
  This will be completed by an evaluation of potential harm, adverse events and safety issues.
Confirm the technical goals of the CCPC platform are met. | From enrollment to the end of follow up at 10 days
  This will be completed via an assessment of the data flow: does the correct patient vitals information reach the clinicians at the right time?
Confirm the technical goals of the CCPC platform are met. | From enrollment to the end of follow up at 10 days
  This will be completed by determining if the CCPC platform provided a holistic view of each patient with vitals, medication, and other collected data.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Pauls Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No